CLINICAL TRIAL: NCT00006391
Title: A Phase I Dose-Finding Study of Oxaliplatin (NSC #266046) Combined With Continuous Infusion Topotecan Hydrochloride as Chemotherapy for Patients With Previously Treated Ovarian Cancer
Brief Title: Oxaliplatin and Topotecan in Treating Patients With Previously Treated Ovarian Epithelial, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068275; U01CA070075 (NIH); P30CA016087 (NIH); NYU-0016; NCI-690
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Oxaliplatin; Topotecan

INTERVENTIONS:
Drug: oxaliplatin
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining oxaliplatin with topotecan in treating patients who have previously treated ovarian epithelial, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxic effects of oxaliplatin and topotecan in patients with previously treated ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the antitumor activity of this treatment regimen in these patients.
* Determine the correlation between the pharmacokinetic and safety data of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oxaliplatin IV over 2 hours on days 1 and 15 and topotecan IV continuously on days 1-15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with measurable disease who achieve a response may receive additional therapy at the discretion of the principal investigator.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin and topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

Patients are followed through day 30.

PROJECTED ACCRUAL: A minimum of 15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer

  * Prior chemotherapy required
* Measurable or evaluable disease
* No symptomatic, untreated brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 4 months

Hematopoietic:

* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) OR
* SGOT no greater than 2.5 times ULN (5 times ULN if liver metastases)

Renal:

* Creatinine no greater than 1.5 times ULN OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No uncontrolled symptomatic congestive heart failure
* No unstable angina pectoris
* No uncontrolled cardiac arrhythmia

Other:

* No other active cancer
* No prior allergy to platinum compounds
* No prior allergic reactions to appropriate antiemetics (e.g., serotonin or antagonists) administered concurrently with study
* No other uncontrolled concurrent illness (e.g., infection)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Chemotherapy
* No concurrent colony stimulating factors during topotecan administration

Chemotherapy:

* See Disease Characteristics
* No prior high-dose chemotherapy requiring bone marrow or peripheral blood stem cell transplantation
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to whole pelvic field
* At least 2 weeks since prior radiotherapy and recovered

Surgery:

* No unresolved sequelae resulting from prior surgery

Other:

* At least 4 weeks since other prior investigational drug
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard S. Hochster, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Hochster H, Chen TT, Lu JM, Hills D, Sorich J, Escalon J, Ivy P, Liebes L, Muggia F. Tolerance and activity of oxaliplatin with protracted topotecan infusion in patients with previously treated ovarian cancer. A phase I study. Gynecol Oncol. 2008 Mar;108(3):500-4. doi: 10.1016/j.ygyno.2007.11.017. Epub 2008 Jan 11. PMID 18191187